CLINICAL TRIAL: NCT05129280
Title: An Open-label, Multicenter, Phase I Study to Evaluate Safety, Pharmacokinetics, and Preliminary Anti-tumor Activity of RO7444973 in Participants With Unresectable and/or Metastatic MAGE-A4-positive Solid Tumors
Brief Title: A Study to Evaluate Safety, Pharmacokinetics, and Preliminary Anti-tumor Activity of RO7444973 in Participants With Unresectable and/or Metastatic MAGE-A4-positive Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to program discontinuation.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BE43244; 2021-000624-35 (EudraCT Number)
Record Dates: First submitted 2021-11-19; First posted 2021-11-22 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I: Single Participant Cohort (SPC) Dose Escalation (Experimental): In Part I, RO7444973 is administered intravenously (IV) every 3 weeks (Q3W) at a fixed dose in a single participant per dose level.
  Interventions: Drug: RO7444973; Drug: Tocilizumab
- Part II: Multiple Participant Cohort (MPC) Dose Escalation (Experimental): In Part II, RO7444973 is administered IV Q3W at a fixed dose in multiple participants per dose level. Step-up dosing may also be explored.
  Interventions: Drug: RO7444973; Drug: Tocilizumab
- Part III: Recommended Phase 2 Dose (RP2D) Expansion (Experimental): Based on emerging data from Part II, an RP2D and dosing regimen will be further investigated in Part III.
  Interventions: Drug: RO7444973; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7444973 — RO7444973 solution for infusion will be administered intravenously at a dose and per schedule as specified for the respective cohort.
Drug: Tocilizumab — Tocilizumab will be used as rescue therapy, in case of clinical presentation of cytokine release syndrome (CRS). Tocilizumab solution for infusion will be administered intravenously at 8 mg/kg for participants >/= 30 kg or at 12 mg/kg for participants < 30 kg.
  Other Names: Actemra, RoActemra

SUMMARY:
This is a first-in-human, open-label, uncontrolled, multi-center, monotherapy dose-escalation and dose expansion study of RO7444973.The aim of this study is to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of RO7444973 in participants with unresectable and/or metastatic melanoma-associated antigen A4 (MAGE-A4)-positive, solid tumors, carrying the HLA-A*02:01 allele.

ELIGIBILITY:
Key Inclusion Criteria:

* Unresectable and/or metastatic solid tumors that have received standard-of-care (SOC) therapies previously and have no other SOC options available
* Confirmed HLA-A*02:01 haplotype
* Confirmed MAGE-A4 expression
* Radiologically measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Life expectancy of >/=12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absence of rapid disease progression, threat to vital organs or non-irradiated lesions >2 cm in diameter at critical sites
* No significant ongoing toxicity from prior anticancer treatment
* Adequate hematological function
* Adequate liver function
* Adequate renal function
* If applicable, willingness to use contraceptive measures.

Key Exclusion Criteria:

* History or clinical evidence of CNS primary tumors or metastases
* Another invasive malignancy in the last 2 years
* Uncontrolled hypertension
* Significant cardiovascular disease
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial, parasitic or other infection
* Current or past history of CNS disease
* Dementia or altered mental status that would prohibit informed consent
* Active auto-immune disease or flare within 6 months prior to start of study treatment
* Expected need for regular immunosuppressive therapy or with systemic corticosteroids
* Insufficient washout from prior anti-cancer therapy
* Prior treatment with a bispecific T-cell engaging or adoptive cell therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From start of treatment up to 90 days after last RO7444973 dose (up to 15 months)
Number of Participants With Dose-limiting Toxicities (DLTs) | From start of treatment up to 21-28 days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From baseline up to 12 months
Disease Control Rate (DCR) | From baseline up to 12 months
Duration of Response (DoR) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 40 months)
Progression-free Survival (PFS) | From baseline to the first occurrence of disease progression or death from any cause, whichever occurs first (up to 40 months)
Overall Survival (OS) | From baseline to death from any cause (up to 40 months)
Pharmacokinetics (PK): Serum Concentration of RO7444973 Over Time | From baseline to end of treatment (EoT) visit within 28 days after the last dose (up to 13 months)
Change from Baseline in Percentage of Participants Positive for Anti-drug Antibodies (ADA) to RO7444973 | From baseline to end of treatment (EoT) visit within 28 days after the last dose (up to 13 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States
- Peter Maccallum Cancer Centre, Melbourne, Victoria, Australia
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Rigshospitalet; Fase 1 Enhed - Onkologi, København Ø, Denmark
- Spain (2):
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitario HM Sanchinarro-CIOCC, Madrid
- Royal Marsden Hospital - Institute of Cancer Research - Sutton, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).